CLINICAL TRIAL: NCT04979286
Title: The Immediate Effect of Gastrocnemius Kinesiotaping on Sprint and Dynamic Balance in Physically Active Children
Brief Title: The Effect of Kinesiotaping on Sprint and Dynamic Balance in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Murat EMİRZEOĞLU, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-44
Record Dates: First submitted 2021-05-04; First posted 2021-07-28 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Sports Performance in Children
Keywords: soccer; child; sprint; dynamic balance; kinesiotaping

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping Group (Experimental): Y strip kinesiotaping will be applied to both the gastrocnemius muscles with approximately 20% tension.
  Interventions: Other: Kinesiotaping
- Placebo Group (Placebo Comparator): Placebo kinesiotaping, approximately 5x5 cm in size, will be applied to the body of both gastrocnemius muscles without any tension.
  Interventions: Other: Placebo Kinesiotaping

INTERVENTIONS:
Other: Kinesiotaping — Y strip kinesiotaping will be applied to both the gastrocnemius muscles while keeping the participant's ankle in full dorsiflexion. The tape will start from the plantar surface of the toe and continue proximally. The medial "Y" tail will be applied along the medial border of the gastrocnemius and the lateral "Y" tail along the lateral border of the gastrocnemius, at approximately 20% tension from the resting length. End points will end just below the popliteal crease.
  Arms: Kinesiotaping Group
Other: Placebo Kinesiotaping — Placebo kinesiotaping, approximately 5x5 cm in size, will be applied to the body of both gastrocnemius muscles without any tension.
  Arms: Placebo Group

SUMMARY:
The aim of this study is to examine the acute effects of kinesio taping applied to the gastrocnemius muscles of children enrolled in soccer school on sprint and dynamic balance.Children who meet the required criteria will be randomly placed in the kinesio taping and placebo groups by drawing lots. Dynamic balance and sprint abilities of the participants were evaluated before and immediately after taping. Y Balance Test will be used to evaluate dynamic balance. Measurements were taken in the anterior, posteromedial and posterolateral directions of the right and left sides.10 m and 20 m sprint tests will be used to assess speed ability. In-group and between-group comparisons will be analyzed using the Statistical Package for the Social Sciences program and appropriate tests.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 8-12
* To be actively participating in football training.

Exclusion Criteria:

* Those with orthopedic, neurological and congenital problems.
* Those with any systematic disease.
* Those who have experience taping before.
* Those who have undergone any surgery within the last 1 year.
* Those who have been absent from training for more than 2 weeks in the last three months.

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
10m Sprint Test | 1 hour
  Sprint
20m Sprint Test | 1 hour
  Sprint
Y-Balance Test | 1 hour
  Dynamic Balance

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)